CLINICAL TRIAL: NCT02046083
Title: Peanut Oral Induction Tolerance in Peanut's Allergic Teenagers
Acronym: PITA 3
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0177; 2013-A00169-36
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Peanut Allergy
Keywords: Teenager; Peanut; OIT (Oral Induction Tolerance)
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- treatment (Experimental): Prospective randomized double blind, placebo controlled, protocol in two phases: 1/ active treatment versus placebo for induction phase; 2/ long versus short maintenance
  Interventions: Drug: arachid
- placebo (Placebo Comparator): Prospective randomized double blind, placebo controlled, protocol in two phases: 1/ active treatment versus placebo for induction phase; 2/ long versus short maintenance

INTERVENTIONS:
Drug: arachid
  Arms: treatment

SUMMARY:
The primary purpose of the protocol is to evaluate the efficacy of a protocol for induction of tolerance to peanut ingestion increasing doses. The secondary purpose is to determine the interest of a prolonged maintenance therapy

DETAILED DESCRIPTION:
Prospective randomized double blind, placebo controlled, protocol in two phases: 1/ active treatment versus placebo for induction phase; 2/ long versus short maintenance

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 12 and 18 years
* Clinical History of allergic manifestation within one hour of ingestion of peanuts or Double-Blind, Placebo-Controlled Food Challenges (DBPCFCs) peanut positive below the threshold of 2 grams
* Bad reaction peanut demonstrated by positive Patch Test (PT ≥ 3 mm above the negative control) and specific IgE f13> 12 IU / mL and / or rAra h2> 5.8 IU / mL
* Previous follow at least 1 year

Exclusion Criteria:

* Lack of response during the initial DBPCFCs to the cumulative dose of 2 grams of peanut or instant dose of 1 gram of peanut
* Uncontrolled asthma and / or severe over the previous year
* Atopic dermatitis uncontrolled
* Initial severe anaphylaxis requiring hospitalization in intensive care
* Presence of a major allergy with anaphylaxis at another allergen risk (milk, egg, nuts, or other)
* Home away from a center could support a severe reaction in emergency
* Lack of motivation and understanding of parents and / or child
* Incapacity

  * to establish a daily logbook of clinical monitoring
  * to support severe reaction after eating peanut
  * to follow a regular peanut ingestion protocol

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients which tolerate the cumulative dose of 2 grams of peanut at the end of the first phase of 24 weeks between treatment and placebo groups | at 24 weeks

SECONDARY OUTCOMES:
Percentage of patients had quadrupled their tolerance to peanut at the end of induction phase | at 24 weeks
Percentage of patients with adverse effects during induction phase | at 24 weeks
Modifications of the immune profile showing a desensitization to peanut | at 24 weeks
Percentage of patients which tolerate the cumulative dose of 2 grams of peanut during a Double-Blind, Placebo-Controlled Food Challenges (DBPCFCs) after 24 weeks without traces eviction diet after the end of maintenance phase | at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc FAUQUERT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Michaud E, Evrard B, Pereira B, Rochette E, Bernard L, Rouzaire PO, Gourdon-Dubois N, Merlin E, Fauquert JL. Peanut oral immunotherapy in adolescents: study protocol for a randomized controlled trial. Trials. 2015 Apr 29;16:197. doi: 10.1186/s13063-015-0717-y. PMID 25925398